CLINICAL TRIAL: NCT04443504
Title: A Pilot Study on the Effectiveness of an Online Intervention for Adoptive Families
Brief Title: An Online Post-Adoption Family Intervention Using Trust-Based Relational Intervention (TBRI) to Improve Understanding, Well-Being, and Connection in Adoptive Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jana Hunsley (Other)
Responsible Party: Sponsor-Investigator, Jana Hunsley, Graduate Research Assistant, Texas Christian University
Organization: Texas Christian University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1920-217
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Family Relations; Parenting
Keywords: post-adoption intervention; Trust-Based Relational Intervention; adoption

STUDY DESIGN:
Intervention Model Description: Two groups will be created using random assignment: an intervention group and a waitlist control group who will receive the intervention 3 months after the intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: The Connected Family Series
- Waitlist Group (No Intervention): The waitlist group will receive the intervention 3 months after the intervention group.

INTERVENTIONS:
Behavioral: The Connected Family Series — The intervention is an online, self-paced post-adoption family intervention that occurs over a 4-week period to support adoptive families post-adoption.
  Arms: Intervention Group

SUMMARY:
The current study aims to examine the effectiveness of an online, self-paced post-adoption intervention to improve understanding, well-being, and connection within adoptive families.To evaluate the effectiveness of this intervention, a mixed method, pre-post design with two conditions will be used. Data from standard, reliable measures and free-response items will be collected pre- and post-intervention from participants in two conditions: the intervention condition and the waitlist condition. The intervention condition involves receiving the intervention immediately following pre-assessments; the waitlist condition involves receiving the intervention approximately 3 months after the intervention condition once all data collection is completed.

The study aims to answer six research questions. Each research question involves analyses of the differences between the intervention and waitlist conditions across multiple time points.

1. What is the intervention's effect on improving awareness of the needs of different family members and understanding how to meet these needs? Hypothesis 1: At post-intervention, parents in the intervention condition will report an improved awareness of the needs of each family member and greater understanding of how to meet these needs.
2. What is the intervention's effect on parent well-being (i.e., parenting confidence and parenting stress) from pre- to post-intervention? Hypothesis 2: Parents in the intervention condition will report increased parenting confidence and trending decreases in parenting stress from pre- to post-intervention compared to those in the waitlist condition.
3. What is the intervention's effect on child well-being (i.e., self-esteem and emotional and behavioral problems) from pre- to post-intervention? Hypothesis 3: Children in the intervention condition will report increased self-esteem and trending decreases in emotional and behavioral problems from pre- to post-intervention compared to those in the waitlist condition.
4. What is the intervention's effect on the quality of the parent-child relationship from pre- to post-intervention? Hypothesis 4: Both parents and children in the intervention condition will report improved connection in the parent-child relationship from pre- to post-intervention compared to those in the waitlist condition.
5. As an exploratory question, what is the intervention's effect on the quality of the sibling relationship from pre- to post-intervention? Hypothesis 5: Children in the intervention condition will report an improvement in the quality of their relationship with their sibling(s) from pre- to post-intervention compared to children in the waitlist condition.
6. What is the intervention's effect on connection and communication within the overall family system from pre- to post-intervention? Hypothesis 6: Parents and children in the intervention condition will report increased family communication and family connection in the whole family system from pre- to post-intervention compared to parents and children in the waitlist condition.

DETAILED DESCRIPTION:
One member of the family will complete a survey to ensure eligibility criteria have been met. In the recruitment application, the individual who completes the application will include an email address to be used as the primary contact person for the family. If the family meets the eligibility criteria, the primary contact person will receive consent forms to complete for each member of the family. Once consent forms are completed for the entire family and each member has agreed to participate in research, the primary contact will complete a demographic survey of basic household information. In the demographic survey, the primary contact will include email addresses for each family member 18 years and older. See timeline below for reference. *Note: dates are approximate.

Once consented, online surveys of pre-assessments will be sent to families via email (via individual links; survey links for children under 18 will be sent to the primary contact). Pre-assessments include individual, dyad, and family measures to examine the effectiveness of the intervention in multiple systems of the family. Each family member who is 12 years and older will complete pre-assessments during a one-week data collection period.

After pre-assessments are complete, families will be randomly assigned to the intervention or waitlist condition using a random number generator, and families will be notified of their assigned condition.

Both the waitlist and intervention condition will complete pre-assessments.

Once the pre-assessment data collection period is complete, families in the intervention condition will have one week before the intervention begins. The primary contact of families assigned to the intervention condition will receive an email with instructions to register and to prepare for the 4-week intervention series. The waitlist condition will do nothing during this time.

One week after pre-assessment data collection is complete, the 4-week intervention series will begin. The intervention includes 4 weekly sessions. Each weekly session involves parents watching a 15-minute mini-webinar, children watching a 5-minute video, parents and children 12 years and older completing separate reflection questions (*note these questions will be used as data for analysis), and families completing two family activities together (an activity aimed at improving connection and an activity aimed at improving communication). The primary contact will complete a checklist of which activities were completed that week. The intervention should take approximately 1.5-3 hours each week for the whole family for a total of 6-12 hours over the 4-week period.

The intervention condition will complete the first week's activities at their own pace within the seven days. On each subsequent Monday of the four weeks, the next week's activities will open for the intervention condition to access. The previous weeks' activities will still be available to the families during the duration of the intervention. All intervention activities will be completed within the four-week time period.

Two weeks after the intervention condition completes the intervention series, post-assessments will be sent to both the intervention and waitlist conditions. Post-assessments will be the same as the pre-assessments in order to examine differences between pre- and post-intervention. Families will have a one-week period to complete the post-assessments.

Three months after the intervention condition completed the intervention, 3-month follow-up assessments will be sent to both the intervention and waitlist conditions. 3-month follow-up assessments will be the same as the pre- and post-assessments. This follow-up data collection period is to determine any longer-term changes that may occur in the family systems post-intervention that may not occur closely following the intervention at the post-intervention data collection time point. Families will have a one-week period to complete the 3-month follow-up assessments.

One week after the three-month follow-up data collection period is completed, families randomly assigned to the waitlist condition will receive the invitation to register for the intervention. The waitlist condition will receive instructions to register for the intervention and to prepare for the 4-week intervention series. The waitlist condition will receive the intervention series in the same order and manner as the intervention condition.

Approximately 6 months after the intervention condition completed the intervention, the intervention condition will complete 6-month follow-up assessments. This follow-up data collection is to determine the long-term changes that may occur in the family system post-intervention. Only the intervention condition will complete this data collection period as the waitlist condition would have completed the intervention at this time.

In total, participation in this study will take approximately 15-20 hours during a 6-month period with approximately 4 hours total to complete surveys and assessments and 6-15 hours to participate in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must be families who have legally adopted or have legal permanency of all children in their family.
* Study participants must have at least one adopted child in the family.
* Adoptive families who have at least two children with at least one child being 12 years or older. It does not matter if the child who is 12 years or older is an adopted or biological child in the family.
* All members of the family must be willing to participate in the intervention and all members 12 years and older must be willing to participate in the research assessments.

Exclusion Criteria:

* Families who are current foster homes.
* Families who have at least one member of the family who has recently been hospitalized for psychiatric issues.
* Families in which at least one member of the family is at risk of harm to self or others.
* Two-parent households in which the marriage is a consistent source of conflict.
* Families who have participated in Hope Connection 2.0, a therapeutic family camp.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Change in Family Cohesion | through study completion, an average of 6 months
  Family Adaptability and Cohesion Scale IV
Change in Parent and Child Relationship | through study completion, an average of 6 months
  Inventory of Parent and Peer Attachment-Revised, Child-Parent Relationship Scale-Short Form

SECONDARY OUTCOMES:
Change in Parenting Stress | through study completion, an average of 6 months
  Parental Stress Scale
Change in Parenting Competence | through study completion, an average of 6 months
  Parenting Sense of Competence Scale
Change in Child Self-Esteem | through study completion, an average of 6 months
  Rosenberg Self-Esteem Scale
Change in Child Emotional and Behavioral Problems | through study completion, an average of 6 months
  Strengths & Difficulties Questionnaire
Change in Sibling Relationship | through study completion, an average of 6 months
  Sibling Relationship Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No